CLINICAL TRIAL: NCT03801499
Title: Lenvatinib for Unresectable Intrahepatic Cholangiocarcinoma: a Single-arm, Phase 2 Trial
Brief Title: Lenvatinib for Unresectable Intrahepatic Cholangiocarcinoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Protocol modification
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Shi Ming, Clinical Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC-S073
Record Dates: First submitted 2019-01-09; First posted 2019-01-11 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Intrahepatic Cholangiocarcinoma
Keywords: Intrahepatic Cholangiocarcinoma; Lenvatinib
MeSH Terms: conditions — Cholangiocarcinoma | interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lenvatinib (Experimental): Participants received lenvatinib capsules 12 milligram (mg) based on the participant's body weight greater than or equal to (>=) 60 kilogram (kg) or 8 mg based on the participant's body weight less than (<) 60 kg at baseline, orally, once daily (QD) up to documented disease progression, development of unacceptable toxicity, participant request, or withdrawal of consent.
  Interventions: Drug: Lenvatinib

INTERVENTIONS:
Drug: Lenvatinib — 12 mg (or 8 mg) once daily (QD) oral dosing.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of lenvatinib for patients with unresectable intrahepatic cholangiocarcinoma

DETAILED DESCRIPTION:
Lenvatinib was non-inferior to sorafenib in overall survival in untreated advanced hepatocellular carcinoma.No study has evaluated the efficacy and safety of lenvatinib in unresectable intrahepatic cholangiocarcinoma. Thus, the investigators carried out this prospective study to find out it.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of unresectable ICC
* Patients must have at least one tumor lesion that can be accurately measured according to mRECIST criteria.
* With no previous treatment
* No Cirrhosis or cirrhotic status of Child-Pugh class A only
* Not amendable to surgical resection ,local ablative therapy and any other cured treatment.
* The following laboratory parameters:

Platelet count ≥ 50,000/μL Hemoglobin ≥ 8.5 g/dL Total bilirubin ≤ 30mmol/ L Serum albumin ≥ 32 g/L ASL and AST ≤ 6 x upper limit of normal Serum creatinine ≤ 1.5 x upper limit of normal INR ≤ 1.5 or PT/APTT within normal limits Absolute neutrophil count (ANC) >1,500/mm3

Exclusion Criteria:

* Evidence of hepatic decompensation including ascites, gastrointestinal bleeding or hepatic encephalopathy
* Known history of HIV
* History of organ allograft
* Known or suspected allergy to the investigational agents or any agent given in association with this trial.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* Evidence of bleeding diathesis.
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.
* Known central nervous system tumors including metastatic brain disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
overall survival (OS) | 12 months
  OS was defined as the duration from the date of randomization until the date of death from any cause. Participants who were lost to follow-up were censored at the last date the participant was known to be alive, and participants who remained alive were censored at the time of data cutoff.

SECONDARY OUTCOMES:
progression free survival (PFS) | 12 months
  PFS was defined as the time from the date of randomization to the date of first documentation of disease progression based on modified Response Evaluation Criteria in Solid Tumors (mRECIST), or date of death, whichever occurred first.
Objective Response Rate (ORR) | 12 months
  ORR was defined as the percentage of participants with a best overall response of complete response (CR) or partial response (PR) based on mRECIST. CR was defined as disappearance of any intratumoral arterial enhancement in all target lesions. PR was defined as at least a 30% decrease in the sum of diameters of viable (enhancement of arterial phase) target lesions taking as reference to the baseline sum of the diameters of target lesions.
Adverse Events | 12 months
  Number of adverse events. Postoperative adverse events were graded based on CTCAE v4.03

CONTACTS AND LOCATIONS:
Overall Officials: Ming Shi, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Cancer Center Sun Yat-sen University, Guangzhou, Guangdong, China